CLINICAL TRIAL: NCT05202847
Title: Pulsed Radiofrequency Ablation to the Modified Ablation Points for Chronic Knee Pain Due to Osteoarthritis: Preliminary Prospective Randomized Controlled Study
Brief Title: Clinial Application of Park et al.(The Knee 27 (2020) 1577-1584)'s Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties in recruiting patients with knee osteoarthritis to the pain clinic.
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji Yeong Kim, Clinical Assistant Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3-2021-0432
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Medical staff performing patient care, including pain management, and investigators who investigate and record observations and evaluations, and participants are kept unaware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulsed radiofrequency ablation to modified points group (Experimental): pulsed radiofrequency ablation aimed at the adjusted target point of Park et al. under C-arm guidance
  Interventions: Procedure: pulsed radiofrequency ablation to modifined points group
- pulsed radiofrequency ablation to conventional points group (Active Comparator): pulsed radiofrequency ablation aimed at conventional target point under C-arm guidance
  Interventions: Procedure: pulsed radiofrequency ablation to conventional points group

INTERVENTIONS:
Procedure: pulsed radiofrequency ablation to modifined points group — Point 1 place 10mm higher than the boundary between Femur's medial epicondyle and shaft. The 2nd point is targeted 20mm above the patella. Point 3 is targeted 10mm above the femur lateral epicondyle and shaft boundary. At point 4, find the boundary position between the tibia epicondyle and the shaft in the AP view and move it superolateral by 10 mm to target the central part of the medial shaft of the tibia and perform the main touch. Point 5 targets the center of the fibular head.
  Arms: pulsed radiofrequency ablation to modified points group
Procedure: pulsed radiofrequency ablation to conventional points group — Under AP view X-ray fluoroscopy, enter the cannula into the tunnel view until reaching the bone, reaching the border of the shaft and epicondyle, then stop the cannula tip at the anterior 2/3 junction in the lateral view. A total of three target points are the boundary position between the femur medial epicondyle and the shaft, the boundary position between the femur lateral epicondyle and the shaft, and the boundary position between the tibia meidal epiconcyle and the shaft. Subsequent procedure will be proceed same as Arm 1
  Arms: pulsed radiofrequency ablation to conventional points group

SUMMARY:
The goal of this study was to perform pulsed radiofrequency ablation with a modified target suggested in the cadaver study by Park et al. (The Knee 27 (2020) 1577-1584) on knee osteoarthritis patients, and to evaluate the effect of reducing the frequency of intravascular injection and reducing pain.

ELIGIBILITY:
Inclusion Criteria:

1. chronic knee pain that does not respond to conservative treatment (physiotherapy, oral analgesic, steroid intra-articular injection, Hyruan injection) for more than 6 months
2. A score of 6 or higher (out of 10) on the target knee's numerical rating scale
3. Knee osteoarthritis 1-4 confirmed in knee X ray within 6 months of study enrollment

Exclusion Criteria:

1. Systemic inflammatory diseases such as rheumatic diseases
2. uncontrolled diabetes
3. malignant tumor
4. If the target knee has a previous surgical history (arthroscopy, arthroscopy, autologous or allograft osteochondral transplantation and autologous cartilage cell transplantation, osteotomy, arthritis surgery)
5. Patients with lidocaine and contrast agent allergy
6. history of nerve block in the target knee within 2 weeks
7. Body mass index over 40 kg/m2
8. bleeding disorder
9. Pregnant/lactating women
10. Inability to understand informed consent and respond to research questionnaires due to cognitive impairment
11. Unable to read consent form (e.g. illiterate, foreigner, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
The rate at which vascular uptake is confirmed when the first contrast agent is given after the needle is positioned at the target point | during the ablation procedure
  Whether vascular uptake is confirmed on the x-ray image is a binary response.

SECONDARY OUTCOMES:
numeric rating score | Before the pulsed radiofrequency ablation, after 4 weeks of the ablaion, after 8 weeks of the ablation, after 12 weeks of the ablation
  A score of 0 indicates no pain and a score of 10 indicates maximum pain.
functional status | Before the pulsed radiofrequency ablation, after 4 weeks of the ablaion, after 8 weeks of the ablation, after 12 weeks of the ablation
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints
quality of life | Before the pulsed radiofrequency ablation, after 4 weeks of the ablaion, after 8 weeks of the ablation, after 12 weeks of the ablation
  Q-5D is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys.
medication | Before the pulsed radiofrequency ablation, after 4 weeks of the ablaion, after 8 weeks of the ablation, after 12 weeks of the ablation
  The Medication Quantification Scale (MQS) is an instrument with potential clinical and research applications for quantifying medication regimen use in chronic pain populations.

IPD SHARING:
Plan to Share IPD: No